CLINICAL TRIAL: NCT05639816
Title: Effect of Common Bile Duct Stone Clearance Using Saline Irrigation After Stone Removal: A Prospective Randomized Control Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 134/2562
Record Dates: First submitted 2022-03-22; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Common Bile Duct Calculi
Keywords: endoscopic retrograde cholangiopancreatography; endoscopic ultrasound; cholangitis
MeSH Terms: conditions — Gallstones; Cholangitis

STUDY DESIGN:
Intervention Model Description: Included patients are randomized to two group, study group and control group an followed up parallelly.
Who Masked: Participant
Masking Description: The patients are blinded to the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- saline irrigation group (Experimental): The patients received saline irrigation of common bile duct after complete ERCP stone removal confirmed by occluded cholangiogram
  Interventions: Procedure: Saline irrigation group
- control (No Intervention): The patients whom complete ERCP stone removal confirmed by occluded cholangiogram were follow up according to standard treatment

INTERVENTIONS:
Procedure: Saline irrigation group — Normal saline irrigation of common bile duct after complete stone removal
  Arms: saline irrigation group

SUMMARY:
Retained CBD stone after ERCP is a common problem in clinical practice. This study aimed to evaluate the effect of saline irrigation of common bile duct after complete stone removal considered by ERCP in the reduction of residual CBD stone and the effect on clinical outcome.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of saline irrigation of common bile duct after complete stone removal considered by ERCP in the reduction of residual CBD stone and the effect on clinical outcome. Patients with CBD stone who received endoscopic stone removal were included after complete stone clearance was seen on occluded cholangiogram. One arm received saline irrigation of CBD at least 50 ml until clear effluent seen and another arm as control. Both group received endoscopic ultrasound to evaluation for residual stone and followed up for complication and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with common bile duct stone
* Complete stone removal by endoscopy as seen in occluded cholangiogram

Exclusion Criteria:

* unstable vital sign
* failed complete stone remval
* assciated biliary malignancy or history of bile duct surgery
* associated bile duct stricture or choledochal cyst
* Toxic cholangitis
* pregnancy or unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
prevalence of residual CBD stone | 1 day
  Detected residual CBD stone by endoscoic ultrasound

SECONDARY OUTCOMES:
factors associated with retained CBD stone | 1 day
  procedural and non-procedural factors related to retained CBD stone
Complicaion and clinical outcome | 6 months
  Complication associated with the procedure, hospital stay, and clinical outcome after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ang TL, Teo EK, Fock KM, Lyn Tan JY. Are there roles for intraductal US and saline solution irrigation in ensuring complete clearance of common bile duct stones? Gastrointest Endosc. 2009 Jun;69(7):1276-81. doi: 10.1016/j.gie.2008.10.018. Epub 2009 Feb 26. PMID 19249039
- [Result] Ahn DW, Lee SH, Paik WH, Song BJ, Park JM, Kim J, Jeong JB, Hwang JH, Ryu JK, Kim YT. Effects of Saline Irrigation of the Bile Duct to Reduce the Rate of Residual Common Bile Duct Stones: A Multicenter, Prospective, Randomized Study. Am J Gastroenterol. 2018 Apr;113(4):548-555. doi: 10.1038/ajg.2018.21. Epub 2018 Mar 27. PMID 29610513